CLINICAL TRIAL: NCT01629121
Title: Prevention of Traumatic Brain Injury in Youth and Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Vernon Barnes, Assistant Professor, Augusta University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GHSF11085
Record Dates: First submitted 2012-06-19; First posted 2012-06-27 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Focus of Study: Bicycle Helmet Wearing Compliance
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- education intervention (Experimental): The intervention delivered education about the benefits of bicycle helmet use and safety and was designed to be sensitive to the age and educational level of the study participant.
  Interventions: Behavioral: education intervention
- control (No Intervention): Printed materials were given to the control group, along with a helmet for each participant.

INTERVENTIONS:
Behavioral: education intervention — The brain injury prevention education intervention included case scenarios as well as education about the benefits of bicycle helmet use. The intervention was designed to be sensitive to the age and educational level of the study participant and his or her parents. Educational materials were chosen to provide use of the five senses to enhance the learning experience. The intervention took place in the privacy of the patient's hospital room. The study was designed so as not to interfere with the hospital standard of care.
  The proper way to fit the bicycle helmet was demonstrated.
  Arms: education intervention

SUMMARY:
The hypothesis was that the implementation of a Safe Kids East Central brain injury prevention program targeting children and caregivers admitted to the Georgia Health Sciences University Children's Medical Center is feasible and that short-term treatment effects of injury prevention education on the child or adolescent and the caregiver will increase bicycle helmet use.

DETAILED DESCRIPTION:
The overarching goal of this project is to reduce traumatic brain injury in children and adolescents by promoting bicycle helmet use via an inpatient educational program. The Safe Kids East Central injury prevention educational program was customized for hospitalized subjects and their caregivers. The investigators hypothesized that this program would increase bicycle helmet use.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in-patients in the Children's Medical Center;
* Projected length of stay >24 hours;
* Mentally and physically fit to complete the educational program;
* History of regular (>1x per week) bicycle riding;
* All racial/ethnic groups.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
parental report of bicycle helmet use | change for baseline in bicycle helmet wearing at 1 and 3 months
  A series of mixed model univariate analyses were used to determine group differences across the follow-ups on helmet wearing.

CONTACTS AND LOCATIONS:
Overall Officials: Vernon A Barnes, PhD, Principal Investigator — Augusta University
Locations (1):
- Georgia Regents University, Children's Medical Center, Augusta, Georgia, United States

REFERENCES:
- [Result] Barnes VA, Maria BL, Caldwell AL, Hopkins I. Prevention of Traumatic Brain Injury in Youth and Adolescents. J Child Neurol. 2013 Nov;28(11):1412-1417. doi: 10.1177/0883073812464272. Epub 2012 Nov 8. PMID 23143720